CLINICAL TRIAL: NCT06577740
Title: Investigation of the Effects of Group-Based and Dual-Task Focused Otago Exercises on Kinesiophobia, Musculoskeletal System and Psychosocial Status in Geriatric Individuals With Kinesiophobia
Brief Title: Group-based and Dual-task Focused Otago Exercises in Geriatric Individuals With Kinesiophobia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Collaborators: Istanbul Gedik University (Other)
Responsible Party: Principal Investigator, ebrar atak, Asst. Prof., Medipol University
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: GroupDualTaskOtagoExercise
Record Dates: First submitted 2024-08-27; First posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Geriatric İndividual Health
Keywords: geriatrics; kinesiophobia; Otago exercises; dual task
MeSH Terms: conditions — Kinesiophobia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Otago Exercise Group (Other): Participants in the study were given group otago exercises for 4 weeks, face to face, once a week for 30 minutes. They were also given brochures containing otago exercises twice a week and followed up remotely. They were asked to walk normally for 30 minutes, 2 days a week. Then they entered a 4-week cleansing period.
  Interventions: Other: Otago Exercise
- Dual Task Focused Otago Exercise Group (Experimental): After a 4-week washout period, participants in the study were given group-based otago exercises and dual-task exercises once a week for 4 weeks. They were given a brochure containing otago exercises including dual-task exercises twice a week and were applied individually and monitored remotely. They were asked to walk normally 2 days a week.
  Interventions: Other: Dual Task Focused Otago Exercise

INTERVENTIONS:
Other: Otago Exercise — Group-based otago exercises were performed for 4 weeks. They were also given a brochure containing otago exercises twice a week and applied individually and followed remotely. They were asked to walk normally for 30 minutes twice a week. They then entered a 4-week washout period.
  Arms: Otago Exercise Group
Other: Dual Task Focused Otago Exercise — After a 4-week washout period, face-to-face group-based and dual-task focused otago exercises were applied once a week for 4 weeks. Participants were given a brochure containing otago exercises including dual-task exercises twice a week and applied individually and monitored remotely. They were asked to walk normally for 30 minutes twice a week.
  Arms: Dual Task Focused Otago Exercise Group

SUMMARY:
The aim of our study was to investigate the effects of group-based and dual-task focused otago exercises on kinesiophobia, musculoskeletal system and psychosocial status in geriatric individuals with kinesiophobia. In the study : 1. Do group-based and dual-task focused otago exercises have an effect on kinesiophobia in geriatric individuals with kinesiophobia? 2. Do group-based and dual-task focused otago exercises have an effect on the musculoskeletal system in geriatric individuals with kinesiophobia? 3. Do group-based and dual-task focused otago exercises have an effect on the psychosocial status of geriatric individuals with kinesiophobia? 4. Do group-based and dual-task focused otago exercises have an effect on cognitive function in geriatric individuals with kinesiophobia? The questions were answered.

DETAILED DESCRIPTION:
Our study was conducted as a cross-controlled study on 20 geriatric individuals. The study lasted 12 weeks. The participants in the study were given group otago exercises for 4 weeks, face to face once a week for 30 minutes, and remotely monitored twice a week with handouts containing the exercises. They were asked to walk normally for 30 minutes on 2 days a week. Then, they entered a 4-week washout period. After the washout period, the participants in the study were given group otago exercises for 4 weeks, face to face for 30 minutes, and remotely monitored twice a week with handouts containing the exercises. They were asked to walk normally for 30 minutes on 2 days a week. Before starting the study, participants were given a demographic information form, Tampa Kinesiophobia Scale for kinesiophobia, Berg Balance Scale for balance assessment, Short Form Geriatric Depression Scale for psychosocial status, 5-times sit-to-stand test to assess fall risk and lower extremity muscle strength, Timed Up and Go test to assess mobility, and Mini Mental State Test and Montreal Cognitive Assessment Test to assess cognitive function. These tests were repeated at the end of the first 4 sessions and the last 4 sessions, and pre- and post-test values were measured.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 65 and over
* Participants who can read and write in Turkish
* Participants who scored 38 or higher on the Tampa Kinesiophobia Scale
* Participants who received 24 points or more from the Mini Mental State Test
* Participating in the study voluntarily
* Individuals who do not have any disability such as vision, hearing, limb loss, etc.
* Participants who can walk independently

Exclusion Criteria:

* Medication status that increases the risk of falls (determined based on information from nursing home nurses and physiotherapists).
* Individuals who are bedridden or wheelchair bound
* Individuals with diagnosed mental or psychological problems (The individual's inability to perceive the scales to be applied)
* Individuals with diagnosed serious neurological or orthopedic problems
* Individuals with diagnosed serious pulmonary or cardiac disease
* Individuals with uncontrolled hypertension or diabetes
* Those with a history of syncope or vertigo attacks in the last 4 weeks

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2024-07-03 (Actual); Study Completion 2024-08-08 (Actual)

PRIMARY OUTCOMES:
Tampa Kinesiophobia Scale | Duration of change in 4 week
  It is a 17-question scale measuring fear of movement/re-injury.
Berg Balance Scale | Duration of change in 4 week
  It is a scale that includes 14 different types of activities aimed at questioning dynamic and static balance.
Geriatric Depression Scale Short Form | Duration of change in 4 week
  It is a scale consisting of 15 questions that determines the level of depression in geriatric individuals.
5 times sit and stand test | Duration of change in 4 week
  Used to assess fall risk and lower extremity muscle strength.
Mini Mental Status Test | Duration of change in 4 week
  It is a scale used to assess cognitive function.
Montreal Cognitive Assessment Test | Duration of change in 4 week
  It is a scale used to identify individuals with mild cognitive impairment and to distinguish them from healthy geriatric individuals.
Timed Up and Go Test | Duration of change in 4 week
  It is a scale used to assess mobility in geriatric individuals.

CONTACTS AND LOCATIONS:
Locations (1):
- Amine Ataç, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It will be evaluated if the researchers are contacted via their e-mail addresses.

REFERENCES:
- [Background] Yang Y, Wang K, Liu H, Qu J, Wang Y, Chen P, Zhang T, Luo J. The impact of Otago exercise programme on the prevention of falls in older adult: A systematic review. Front Public Health. 2022 Oct 20;10:953593. doi: 10.3389/fpubh.2022.953593. eCollection 2022. PMID 36339194